CLINICAL TRIAL: NCT01170039
Title: A Randomized, Double Blind, Placebo-controlled Trial to Examine the Effectiveness of Lubiprostone on Constipation Symptoms and Colon Transit Time in Diabetic Patients
Brief Title: The Effectiveness of Lubiprostone in Constipated Diabetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jennifer Christie, MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00014592
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Constipation; Diabetes
Keywords: Constipation; Diabetes; Lubiprostone; Amitiza; African Americans
MeSH Terms: conditions — Constipation; Diabetes Mellitus | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone (Active Comparator)
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — Lubiprostone will be given as 24 mcg orally twice a day.
  Other Names: Amitiza
  Arms: Lubiprostone
Drug: Placebo — A matched placebo pill will be given twice a day for 8 weeks.
  Arms: Placebo

SUMMARY:
The investigators will recruit a total of 136 diabetic men and women with constipation into this study from both The Emory Clinic and The Atlanta Veteran's Administration Hospital. The investigators will track spontaneous bowel movements defined as a bowel movement in 24 hours after initiation of study drug (SBMs) in all patients two weeks before treatment with lubiprostone as well as measure baseline colonic transit using the Smartpill pH capsule. Colon transit reflects that rate of colonic peristalsis and movement of stool through the large bowel.

Patients will receive either lubiprostone 24 micrograms (mcg) orally twice a day for 8 weeks or placebo. Primary and secondary endpoints will be the number of SBMs/week and colonic transit time as measured by the Smartpill capsule, respectively. The number of SBMs/week will be evaluated at 0, 2, 4 and 8 weeks after initiation of therapy. The investigators will over-sample African American patients to achieve approximately 50% enrollment of this group. In a subanalysis, the investigators will assess response to treatment between the general population and African Americans.

We hypothesize that lubiprostone will significantly increase the number of SBMs as well as decrease colonic transit time and improve quality of life in constipated diabetic patients compared with placebo.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is very common in the United States, and the incidence as well as prevalence of this disease are increasing. DM is not only a risk factor for cardiovascular and pulmonary conditions, but is also linked with several digestive complications. Among digestive complaints, constipation occurs in approximated two-thirds of patients with DM, making constipation the most common gastrointestinal (GI) complaint among type 2 diabetics. Consequently, these patients suffer abdominal pain, bloating, and have a lower health related quality of life when compared with patients without DM and GI symptoms.Constipated individuals may be reluctant to eat on a regular schedule which may worsen glycemic control as well as the symptoms related to an underlying diabetic enteropathy.

Effective therapies for constipation are limited and there is little data evaluating the treatment of constipation, specifically in diabetic patients. Lubiprostone has been shown to be superior to placebo in increasing the number of spontaneous bowel movements (SBMs) in patients with chronic idiopathic constipation (CIC) and irritable bowel syndrome with constipation (IBS-C). However, lubiprostone has not been previously studied in diabetics suffering with constipation. Furthermore, other prokinetic pharmacotherapeutics targeted toward constipated patients with diabetes mellitus type 2 are lacking.

African Americans have the highest rate of DM compared with other ethnic groups in the Unites States. Furthermore, constipation is more prevalent in African Americans compared with other minority groups. However, there is little data evaluating the prevalence of constipation and the response to treatment in African Americans. Therefore, more information regarding the severity of symptoms, differences in bowel patterns, colonic transit, and response to therapy is important to improving the management of constipation in this group. Hence, in a subanalysis, we will study whether the responsiveness of African American patients to lubiprostone differs from that of the general population.

Given the dearth of information on the effectiveness of lubiprostone in diabetics, who have a particularly strong need for alternative safe and effective treatments for constipation, we propose to assess the effectiveness of lubiprostone in constipated diabetic men and women.

This is a randomized double- blind placebo controlled trial of lubiprostone in the treatment of constipation in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with constipation.
* Patient must be on stable oral or subcutaneous hypoglycemic medication for 6 months.

Exclusion Criteria:

* Acute infections
* Ischemic bowel syndrome
* Gastrointestinal obstruction

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Christie, MD, Principal Investigator — Emory University; Latoya Carter, Study Director — Emory University
Locations (2):
- United States (2):
  - Atlanta Veterans Administration Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from The Emory Clinic and The Atlanta Veterans Administration Hospital from August 2011 to September 2014.
Pre-assignment Details: 121 subjects were enrolled in the study; there were 4 Screen Failures, 22 drop outs prior to randomization and 19 subjects were Early Terminations. 76 subjects were randomized and underwent a two-week wash-out period during which they did not take any laxatives.
Groups:
- Lubiprostone: Subjects with diabetes and constipation received 24 mcg of lubiprostone orally twice a day for 8 weeks.
- Placebo: Subjects with diabetes and constipation received a placebo pill twice a day for 8 weeks.
Period: Overall Study
Arm/Group | Lubiprostone | Placebo
Started | 37 | 39
Completed | 29 | 33
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lack of funding, drug not available | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone | Placebo | Total
Number analyzed (Participants) | 37 | 39 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 39 | 76
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States | 37 | 39 | 76

OUTCOME MEASURES:

1. Primary Outcome: Efficacy, Measured by the Average Number of Spontaneous Bowel Movements (SBMs) Per Week
Description: The average number of spontaneous bowel movements calculated per week from baseline to 8 weeks was recorded. The number of spontaneous bowel movements was recorded by the subjects in a daily stool diary and the weekly average was calculated. Spontaneous bowel movements are bowel movements within a 24 hour period independent of rescue medication use within the previous week.
Time Frame: 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks
Population: Two subjects in the Lubiprostone arm did not complete the daily stool diary at baseline. No data was analyzed for these two subjects.
Measure: Mean (Standard Deviation); unit: spontaneous bowel movements
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 35 | 39
spontaneous bowel movements
  1 week | 4.85 (5.27) | 1.40 (3.27)
  2 weeks | 3.81 (5.60) | 2.41 (4.29)
  3 weeks | 5.76 (4.99) | 3.11 (4.34)
  4 weeks | 4.12 (4.63) | 2.48 (3.68)
  5 weeks | 5.28 (4.10) | 3.03 (4.33)
  6 weeks | 4.52 (5.37) | 3.23 (3.95)
  7 weeks | 4.65 (5.27) | 3.46 (3.59)
  8 weeks | 5.30 (4.42) | 2.63 (3.81)

2. Secondary Outcome: Efficacy, Measured by the Duration of Colonic Transit Time as Measured by the SmartPill pH Capsule
Description: The duration of colonic transit time in hours was measured by the SmartPill pH Capsule. Colonic transit time is the time interval from the cecal entry of the capsule to anal expulsion and was measured in hours.
Time Frame: Baseline, 4 weeks
Population: Intention to treat population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 37 | 39
hours
  Baseline n=30; n=32 | 45.3 (25.7) | 40.9 (28.6)
  4 weeks n=24; n=22 | 36.2 (28.1) | 47.7 (27.7)

3. Secondary Outcome: Number of Subjects With Daily Abdominal Discomfort
Description: The number of subjects experiencing abdominal discomfort was recorded weekly.
Time Frame: 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks
Population: The number of participants in both arms was analyzed by Intention-to-Treat (ITT).
Measure: Number; unit: participants
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 37 | 39
participants
  1 week (n=33; n=38) | 24 | 26
  2 weeks (n=32; n=37) | 17 | 20
  3 weeks (n=29; n=33) | 17 | 21
  4 weeks (n=30; n=33) | 16 | 22
  5 weeks (n=27; n=33) | 13 | 18
  6 weeks (n=26; n=30) | 20 | 14
  7 weeks (n=23; n=29) | 14 | 16
  8 weeks (n=22; n=29) | 11 | 15

4. Secondary Outcome: Change in Scores on the Patient Assessment of Constipation Quality of Life (PAC-QOL) Questionnaire
Description: The difference in the scores on the self-reported Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaire. The quality of life is measured by the by the overall scores on the Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaire, a validated 28-item questionnaire measuring quality of life as it pertains to constipation. The 28 items are grouped into four subscales, 1) worries and concerns, 2) physical discomfort, 3) psychosocial discomfort, and 4) satisfaction. A 5-point Likert response scale, ranging from 0 (Not at all/None of the time) to 4 (Extremely/ All of the time), is used. The subscale scores vary from 0 to 4 and the total (global) score ranges from 0 to 4. A lower score indicates better quality of life (QOL).
Time Frame: Screening, 8 weeks
Population: 7 subjects in the Lubiprostone arm and 7 subjects in the placebo arm did not complete the Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaire and therefore no data was analyzed for these subjects.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 30 | 32
scores on a scale
  Global Score | -0.91 (0.64) | 1.19 (1.07)
  Physical discomfort | -1.08 (0.71) | -1.22 (1.05)
  Psychosocial discomfort | -0.72 (0.72) | -1.13 (1.07)
  Worries and concerns | -0.88 (0.79) | -1.18 (1.29)
  Satisfaction | -1.28 (1.28) | -1.26 (1.43)

ADVERSE EVENTS:
Arm/Group | Lubiprostone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/39
Other Adverse Events (participants affected / at risk) | 28/37 | 25/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lubiprostone (N=37) | Placebo (N=39)
Nausea (Gastrointestinal disorders) | 15 | 9
Bloating (Gastrointestinal disorders) | 14 | 11
Diarrhea (Gastrointestinal disorders) | 12 | 3
Abdominal Pain (Gastrointestinal disorders) | 11 | 8
Vomiting (Gastrointestinal disorders) | 3 | 2
Headache (Nervous system disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes